CLINICAL TRIAL: NCT03097471
Title: Prospektive, Klinische Studie Zur Marktbeobachtung (Post Market Follow-Up Study) Der Knieendoprothese BPK-S Integration Aus Keramikwerkstoff BIOLOX (R) Delta (Prospective Clinical Post Market Follow-up Study of the Total Knee Endoprosthesis BPK-S (Brehm Precision Knee System)Made of Ceramic Material BIOLOX (R) Delta
Brief Title: BPK-S Integration (Ceramic) Post Market Clinical Follow-Up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Klemens Trieb (Other)
Responsible Party: Sponsor-Investigator, Klemens Trieb, Univ. Prof. Dr. Klemens Trieb, Klinikum Wels-Grieskirchen
Organization: Klinikum Wels-Grieskirchen (Other)
Other Study IDs: BPK-S-(pKK)-01-2011
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Restoration if Knee Joint Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BPK-S Integration (Ceramic) — primary total knee endoprosthesis

SUMMARY:
Post-market prospective clinical study with a medical device. Data from patients that routinely receive a primary BPK-S-integration knee implant made of ceramic will be documented with a follow-up time of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Congenital or acquired knee joint defects/deformation which necessitate the implantation of a knee joint replacement
* Defects or malfunctions of the knee joint
* Degenerative, rheumatic, post-traumatic arthritis/arthrosis
* Symptomatic knee instability
* Reconstruction of flexibility
* Patients with material hypersensitivity

Exclusion Criteria:

* Obesity or overweight of the patient
* Acute or chronic infections near the implantation
* Diseases that impair bone growth such as cancer, renal dialysis, osteopenia, etc.
* Sensitivity to foreign matter in the implant materials
* Bone tumors in the area of the implant anchoring
* Illnesses which can be treated without using a knee implant
* Lack of patient cooperation
* Abuse of medication, drug abuse, alcoholism or mental disease
* Pregnancy
* Serious osteoporosis
* Serious damage to the bone and soft tissue structures which impedes stable anchoring and joint function
* Systemic diseases and metabolic disorders
* Overload of the knee implant to be expected

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who routinely receive an BKP-S Integration implant made of ceramic are asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Improvement of Knee Society Score | 12 months

SECONDARY OUTCOMES:
Improvement of Knee Society Score over the course of the study | 3 months, 24 months
Improvement of EQ-5D (Euroquol 5 dimension) score | 3 month, 12 months, 24 months
Improvement of Oxford Score | 3 month, 12 months, 24 months
Documentation of Complications | 3 month, 12 months, 24 months

IPD SHARING:
Plan to Share IPD: No